CLINICAL TRIAL: NCT02795637
Title: Pharmacokinetics of Orally Administered Dasotraline in Subjects With Mild, Moderate, and Severe Hepatic Dysfunction
Brief Title: Study of the What the Body Does to the Drug in Subjects With Mild, Moderate, and Severe Liver Dysfunction
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sumitomo Pharma America, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SEP360-103
Record Dates: First submitted 2016-05-23; First posted 2016-06-10 (Estimated); Last update posted 2016-12-02 (Estimated); Status verified 2016-12

CONDITIONS: Attention Deficit Hyperactivity Disorder (ADHD); Binge-Eating Disorder Disorder
Keywords: Attention deficit hyperactivity disorder (ADHD),; Binge-Eating Disorder (BED)
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity; Binge-Eating Disorder | interventions — 4-(3,4-dichlorophenyl)-1,2,3,4-tetrahydronaphthalen-1-amine; SEP 225289

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- dasotraline (Experimental): dasotraline 8mg capsule/day
  Interventions: Drug: dasotraline

INTERVENTIONS:
Drug: dasotraline — dasotraline 8mg capsule/day
  Other Names: SEP225289

SUMMARY:
Study of the what the body does to the drug in subjects with mild, moderate, and sever liver dysfunction (not working properly)

DETAILED DESCRIPTION:
This is an open-label single-dose study. Approximately 40 total subjects will be enrolled. In each of the 3 hepatic impairment groups (mild hepatic dysfunction [Child-Pugh score of 5 - 6], moderate hepatic dysfunction [Child-Pugh score of 7 - 9], severe hepatic dysfunction [Child Pugh score of 10 - 12]) approximately 10 subjects will be enrolled in order to achieve 8 subjects completing the study in each group. In addition, approximately 8 12 healthy subjects with non-impaired hepatic function will be enrolled to match the subjects in the hepatic impairment groups. Subjects with non-impaired hepatic function may be matched to more than 1 hepatically impaired subject and may be matched to impaired subjects in different Child-Pugh categories; ie, mild, moderate, and/or severe. In order to obtain matched control subjects, after each subject with hepatic impairment has completed the study, a subject with non-impaired hepatic function will be sought; the already enrolled matched control subjects will be checked for a match prior to screening and enrollment of a new match. Each matched control subject will be selected to be demographically comparable to one or more hepatic dysfunction subjects in age (± 10 years), gender, and weight (± 20%). Subjects who do not complete the study may be replaced in order to achieve 8 subjects completing the study in each hepatic impairment group and appropriate healthy matched control subjects.

The study will consist of Screening (Days -28 to -2), Inpatient Period (Days 1 through 7), and Follow-up (Days 8 28). Screening assessments will be used to classify the degree of a subject's hepatic impairment. The degree of impairment will be assigned based on the Child-Pugh category for classification for severity of liver disease. Subjects will be admitted to the clinical site on the day prior to administration of study drug and remain inpatient until discharge on Day 7 (approximately 168 hours after treatment). Subjects may be discharged on Day 5, if in the investigator's opinion they can be relied upon to return for the Day 6 and 7 visits. The following safety assessments will be performed: physical examination; vital signs; clinical laboratory evaluations (hematology, prothrombin time, serum chemistry, and urinalysis); AE collection, ECGs, and C SSRS. Blood and urine samples will be collected for analyses of study drug concentrations and plasma protein binding. The blood sampling duration (648 hours postdose [Day 28]) was chosen to determine the terminal half-life of dasotraline, with the expectation that this time may be extended in hepatically impaired subjects compared to the control subjects. A blood sample for pharmacogenetics will be collected only from subjects who provide separate informed consent to collect this sample. The sample will be utilized for potential evaluation of genetic polymorphisms upon selected enzymatic pathway(s) responsible for the metabolism of dasotraline; this sample is optional for participation in the study.

Exclusion Criteria continued from Eligibility Section:

Any subject with hepatic impairment meeting any of the following criteria will be excluded:

1. Subject who does not tolerate venipuncture or has poor venous access that would cause difficulty for collecting blood samples.
2. Subject with a Child-Pugh classification score ≥ 13.
3. Subject with encephalopathy grade > 1.
4. Subject experienced hepatic coma within the 12 months prior to screening.
5. Subject, who has any abnormal medical history, physical examination, ECG, or laboratory result which, in the opinion of the investigator and medical monitor, may affect the safety of the subject. Subjects with abnormal medical history that is stable may be enrolled.
6. Subject with clinically significant cardiovascular disease, including any of the following:

   1. history of cardiac surgery or myocardial infarction within 6 months prior to screening;
   2. unstable coronary artery disease;
   3. congestive heart failure greater than New York Heart Association (NHYA) Functional Class 1;
   4. cardiac arrhythmia or conduction disturbance resulting in atrioventricular block (AV) block, ventricular fibrillation or causing syncope, near syncope or other alterations of mental status;
   5. severe mitral or aortic valvular disease;
   6. moderately symptomatic peripheral vascular disorder;
   7. uncontrolled hypertension (systolic blood pressure > 200 mmHg and/or diastolic blood pressure > 110 mmHg). However, subjects with stable mild hypertension who are controlled with the same medication over the 2 months prior to screening may be enrolled in the study.
   8. any other cardiovascular condition which, in the opinion of the investigator or medical monitor, might interfere with the results or conduct of the study.
7. Subject has had hepatic transplant or has systemic lupus erythematosus or hepatic carcinoma, or is on the liver transplant list.
8. Subject has estimated creatinine clearance ≤ 60 mL/min according to the Cockcroft-Gault equation.
9. Subject with therapeutic paracentesis within 15 days prior to administration of study drug.
10. Subject has had an acute illness within 30 days prior to administration of study drug.
11. Subject who has had a febrile illness within 14 days prior to administration of study drug.
12. Subject has a disorder or history of a condition that may interfere with drug absorption, distribution, metabolism or excretion including clinically significant abnormality of the renal system, a history of malabsorption, or previous gastrointestinal surgery that could affect drug absorption or metabolism.
13. Subject has a presence or history of any medically diagnosed, clinically significant psychiatric disorder (including intellectual disability and substance-related disorders). Note: For subject with a history of substance-related disorder or alcohol related disorder as defined by DSM 5 criteria the condition must have been more than 1 year prior to screening.
14. Subject has an average weekly alcohol intake that exceeds 21 units per week (males up to age 65) and 14 units per week (males over age 65 and females). 1 unit = 12 oz or 360 mL or beer; 5oz or 150 mL of wine; 1.5 oz or 45 mL of distilled spirits.
15. Subject is unwilling to stop alcohol consumption for at least 48 hours prior to admission on Day -1 (as confirmed by breath or urine alcohol test) through Day 7.
16. Subject has had a portal systemic shunt including portal-systemic shunts (PSS) and transjugular I ntrahepatic portosystemic shunt (TIPS).
17. Subject has shown evidence of hepatorenal syndrome.
18. Subject has required treatment for gastrointestinal bleeding or encephalopathy within the 12 months prior to screening.
19. Subject has had significant blood loss (> 500 mL) or donated blood, plasma, or other blood products within 30 days prior to administration of study drug.
20. Subject with known significant bleeding diathesis, which could preclude multiple venipunctures (for example, history of recent bleeding from esophageal varices, or platelet count less than 40,000/microliters or hemoglobin < 10 g/dL).
21. Subject has exhibited evidence of acute viral hepatitis between the start of screening and study drug administration.
22. Subject answers "yes" to "Suicidal Ideation" Items 4 or 5 on the C SSRS. Subjects who have significant findings for suicidal ideation upon completion of the C SSRS must be referred to the investigator for follow-up evaluation.
23. Subject tests positive at screening for the HIV 1 or HIV 2 antibody.
24. Subject has a positive urine alcohol test.
25. Subject with albumin, potassium, magnesium and/or calcium outside the normal limits of the reference range may be included at the investigator's discretion.
26. Subject has used any drugs known or suspected to affect hepatic or renal clearance capacity within 30 days prior to administration of study drug.
27. Subject has taken any prescription or OTC medications, herbal tea, energy drinks, herbal products (eg, St John's Wort, milk thistle, etc) or supplement/supra-therapeutic doses of vitamins within 5 half lives or 14 days (whichever is longer) prior to administration of study drug or is anticipated to need any medication during the study, with the exception of those permitted by the protocol or approved by the investigator and medical monitor. Note: All drugs will be reviewed on a case-by-case basis by the medical monitor and are prohibited unless deemed acceptable by the investigator and medical monitor.
28. Subject who has previously received dasotraline.
29. Subject has history of intolerance to stimulants.
30. Subject has a history of allergic reaction or has a known or suspected sensitivity to any substance that is contained in the study drug formulation.
31. Subject has taken any investigational drug within 30 days or 5 half lives (whichever is longer) prior to administration of study drug.
32. Subject is currently a heavy user of nicotine, ie, smoking more than 20 cigarettes (eg, 1 pack) per day or equivalent (eg, e-vapor cigarette, pipe, cigar, chewing tobacco, nicotine patch or nicotine gum).
33. Subject cannot comply with the smoking restrictions of the study site during the confinement period or is unable or unwilling to refrain from smoking and tobacco use for 2 hours prior to study drug administration and 4 hours following administration.
34. Subject has a need for special dietary restrictions, unless the restrictions are approved by the investigator and medical monitor.
35. Subject with a history or suspicion of barbiturate, amphetamine, or narcotic abuse and/or positive screening result for any of these substances. Subjects who are currently receiving prescription narcotic pain relievers may be included at the investigator's and medical monitor's discretion.
36. Subject who received live vaccine(s) within 1 month prior to screening, or intends to during the study. Note: Influenza vaccine will be allowed, if administered > 21 days prior to study drug administration.

ELIGIBILITY:
Inclusion Criteria:

Subjects with non-impaired hepatic function must meet all of the following criteria:

1. Male or nonpregnant, nonlactating female between 18 and 70 years of age.
2. Subject must have a normal neurologic exam including tests for impending hepatic encephalopathy.
3. Subject's weight is at least 50 kg.
4. Subject's body mass index (BMI) is at least 18 kg/m2 but no more than 37 kg/m2
5. Subject must be in general good health be demographically comparable to a least 1 subject with hepatic impairment who completed the study.
6. Subject has a negative urine drug screen (UDS).

Subjects with hepatic impairment must meet all of the following criteria:

1. Male or nonpregnant, nonlactating female between 18 and 70 years of age.
2. Subject must have a normal neurologic exam including tests for impending hepatic encephalopathy. Note: Subjects with grade 0 or 1 hepatic encephalopathy will be considered for enrollment in the study.
3. Subject's weight is at least 50 kg.
4. Subject's BMI is at least 18 kg/m2 but no more than 37 kg/
5. Subject has a negative UDS.
6. Subject with stable, chronic medical conditions (eg, hypertension and hyperlipidemia) in addition to hepatic impairment that, in the opinion of the investigator, will not significantly alter the disposition of the study drug, will not place the subject at increased risk by participating in the study, and will not interfere with interpretation of the data may be permitted to enroll in the study after discussion and agreement between the investigator and medical monitor.
7. Subject exhibits vital signs within the reference range for their age and level of hepatic impairment; subjects with vital signs outside the reference ranges may be eligible for the study if the investigator and medical monitor agree that the results are not clinically significant based on the age and hepatic impairment status of the subject, and will not impact study conduct.
8. Subject with out-of-range laboratory results that are related to the subject's underlying condition are eligible; however, the results will need to be carefully reviewed by the investigator and medical monitor to determine if a subject is eligible for study participation. Out of range results could indicate a stable or unstable situation. If the subject is unstable (eg, rapidly changing liver tests, significantly worsened anemia compared to earlier labs, etc), then such subject would be excluded from study participation. Serum bilirubin, albumin, and prothrombin time will be assessed individually for a point score according to the Child-Pugh classification.
9. Subject has a diagnosis of chronic hepatic impairment for at least 6 months and, in the opinion of the investigator, the severity of the subject's hepatic disease is stable, which is defined as having no clinically significant change in disease status within the 90 days prior to study drug administration, as documented by the subject's recent medical history. Copies of documentation of any clinical information used to make a previous diagnosis of hepatic dysfunction must be available. This may include abnormal liver function tests, clinical evidence of portal hypertension, a positive liver biopsy (eg, for cirrhotic disease, portal hypertension), and/or hepatic ultrasound.
10. The total score of the Child Pugh classification must be 5 or 6 for subjects with mild hepatic dysfunction, and between 7 and 9, inclusive, for subjects with moderate dysfunction, and between 10 and 12, inclusive, for subjects with severe hepatic dysfunction.
11. Subject receiving medication for underlying disease states or medical conditions related to hepatic dysfunction must be on a stable dose of medication and/or treatment regimen. Subjects who are receiving a fluctuating treatment regimen may be considered for inclusion if, in the opinion of the investigator, the underlying disease is under control; however these subjects must have medical monitor approval.
12. Subject with a history of hepatic impairment due to hepatitis B is eligible provided there is no evidence of an active disease state, defined as a positive hepatitis B antigen test at screening.
13. Subject with a history of alcohol abuse is eligible provided the urine alcohol test is negative.
14. Subject with a history of type 2 diabetes mellitus is eligible provided that, in the investigator's opinion, he or she has stable diabetes.

Exclusion Criteria:

Any subject with non-impaired hepatic function meeting any of the following criteria will be excluded:

1. Subject who does not tolerate venipuncture or has poor venous access that would cause difficulty for collecting blood samples.
2. Subject has any clinically significant unstable medical abnormality, chronic disease, or history of clinically significant abnormality of the cardiovascular, respiratory, hepatic or renal systems.
3. Subject has any clinically significant abnormal medical history, physical examination, ECG, or laboratory results.
4. Subject has estimated creatinine clearance ≤ 60 mL/min according to the Cockcroft Gault equation.
5. Subject has had an acute illness within 30 days prior to administration of study drug.
6. Subject who, within 14 days prior to administration of study drug, has had a febrile illness.
7. Subject has a disorder or history of a condition that may interfere with drug absorption, distribution, metabolism or excretion including clinically significant abnormality of the hepatic or renal system, a history of malabsorption, or previous gastrointestinal surgery that could affect drug absorption or metabolism.
8. Subject has a presence or history of any medically diagnosed, clinically significant psychiatric disorder (including intellectual disability and substance-related disorders).
9. Subject answers "yes" to "Suicidal Ideation" Items 4 or 5 on the C SSRS. Subjects who have significant findings for suicidal ideation upon completion of the C SSRS must be referred to the investigator for follow-up evaluation.
10. Female subject who is pregnant, lactating, or within 6 months postpartum.
11. Subject tests positive at screening for the hepatitis B surface antigen or hepatitis C antibody or human immunodeficiency virus (HIV 1 or HIV 2) antibody.
12. Subject has a positive urine alcohol test.
13. Subject has history of substance-related disorder or alcohol related disorder as defined by Diagnostic and Statistical Manual of Mental Disorders, 5th Edition (DSM 5) criteria within 1 year prior to screening.
14. Subject has an average weekly alcohol intake that exceeds 21 units per week (males up to age 65) and 14 units per week (males over age 65 and females). 1 unit = 12 oz or 360 mL of beer; 5 oz or 150 mL of wine; 1.5 oz or 45 mL of distilled spirits.
15. Subject is unwilling to stop alcohol consumption for at least 4 hours prior to admission on Day -1 (as confirmed by breath or urine alcohol test) through Day 7.
16. Subject who has previously received dasotraline.
17. Subject has history of intolerance to stimulants.
18. Subject has history of allergic reaction or has a known or suspected sensitivity to any substance that is contained in the study drug formulation.
19. Subject has had significant blood loss (> 500 mL) or donated blood, plasma, or other blood products within 30 days prior to administration of study drug.
20. Subject has used any drugs known or suspected to affect hepatic or renal clearance capacity within 30 days prior to administration of study drug.
21. Subject has taken any prescription or over-the-counter (OTC) medications, herbal tea, energy drinks, herbal products (eg, St John's Wort, milk thistle, etc) or supplement/supra-therapeutic doses of vitamins within 5 half lives or 14 days (whichever is longer) prior to administration of study drug or is anticipated to need any medication during the study, with the exception of those permitted by the protocol or approved by the investigator and medical monitor.
22. Subject has taken any investigational drug within 30 days or 5 half lives (whichever is longer) prior to administration of study drug.
23. Subject is currently a heavy user of nicotine, ie, smoking more than 20 cigarettes (eg, 1 pack) per day or equivalent (eg, e-vapor cigarette, pipe, cigar, chewing tobacco, nicotine patch or nicotine gum).
24. Subject cannot comply with the smoking restrictions of the study site during the confinement period or is unable or unwilling to refrain from smoking and tobacco use for 2 hours prior to study drug administration and 4 hours following administration.
25. Subject with history or suspicion of barbiturate, amphetamine, or narcotic abuse and/or positive screening results for any of these substances. Subjects who are currently receiving prescription narcotic pain relievers may be included at the investigator's and medical monitor's discretion.
26. Subject who received anticoagulant therapy within 90 days prior to administration of study drug.

27 Subject who received live vaccine(s) within 1 month prior to screening, or intends to during the study. Note: Influenza vaccine will be allowed, if administered > 21 days prior to study drug administration.

28. Subject has used a strong inhibitor or inducer of cytochrome P450 enzymes within 30 days prior to admission.

Please see additional eligibility criteria in the Study Description section, under Detailed Description

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2016-05; Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Plasma PK parameters: Area under the plasma/serum concentration-time curve from time zero to infinity (AUC0 inf) | Day 1 -28
  Plasma PK parameters: Area under the plasma/serum concentration-time curve from time zero to infinity (AUC0 inf)
Plasma PK parameters: time of occurrence of Cmax | Day 1 -28
  Plasma PK parameters: time of occurrence of Cmax

SECONDARY OUTCOMES:
Urine PK parameters: amount excreted in urine from time zero to time t (AEx0 t) | Day 1 -28
  Urine PK parameters: amount excreted in urine from time zero to time t (AEx0 t)
Urine PK parameters: renal clearance (CLR) | Day 1 -28
  Urine PK parameters: renal clearance (CLR)
Urine PK parameters: percent of dose excreted in urine (%fe) | Day 1 -28
  Urine PK parameters: percent of dose excreted in urine (%fe)
Unbound fraction of dasotraline in plasma at 10, 12, and 24 hours postdose . | 0-24 hours
  Unbound fraction of dasotraline in plasma at 10, 12, and 24 hours postdose .
Incidence of adverse events (AEs), SAEs, and AEs resulting in study discontinuation. | Day 1 -28
  Incidence of adverse events (AEs), SAEs, and AEs resulting in study discontinuation.
Absolute values and changes from baseline in clinical laboratory tests (hematology, serum chemistry, urinalysis, prothrombin time), vital signs (respiratory rate, body temperature, supine blood pressure, and supine pulse rate), and 12 lead ECGs. | Day 1 to 28
  Absolute values and changes from baseline in clinical laboratory tests (hematology, serum chemistry, urinalysis, prothrombin time), vital signs (respiratory rate, body temperature, supine blood pressure, and supine pulse rate), and 12 lead ECGs.
Frequency of subjects with suicidal ideation or suicidal behavior using the Columbia Suicide Severity Rating Scale (C SSRS). | Day 1 to 28
  Frequency of subjects with suicidal ideation or suicidal behavior using the Columbia Suicide Severity Rating Scale (C SSRS).
Plasma PK parameters: AUC0-last, area under the blood concentration time curve from time zero to 24 hours postdose (AUC0-24) | Day 1 - 28
  Plasma PK parameters: AUC0-last, area under the blood concentration time curve from time zero to 24 hours postdose (AUC0-24)
Plasma PK parameters: t1/2 | Day 1 - 28
  Plasma PK parameters: t1/2
Plasma PK parameters: lag time (tlag) | Day 1 - 28
  Plasma PK parameters: lag time (tlag)
Plasma PK parameters: time of occurrence of Cmax (tmax) | Day 1 -28
  Plasma PK parameters: time of occurrence of Cmax (tmax)
Plasma PK parameters: apparent clearance (CL/F) | Day 1 - 28
  Plasma PK parameters: apparent clearance (CL/F)
Plasma PK parameters: apparent volume of distribution (Vz/F) | Day 1 - 28
  Plasma PK parameters: apparent volume of distribution (Vz/F)

CONTACTS AND LOCATIONS:
Overall Officials: CNS Medical Director, Study Director — Sumitomo Pharma America, Inc.
Locations (5):
- United States (5):
  - Clinical Pharmacology of Miami, Inc., Miami, Florida
  - Orlando Clinical Research Center, Orlando, Florida
  - Atlanta Center for Medical Research, Atlanta, Georgia
  - DaVita Clinical Research, Minneapolis, Minnesota
  - American Research Cororation (ARC), Texas Liver Instituete (TLI), San Antonio, Texas